CLINICAL TRIAL: NCT01793415
Title: Phase 1 + 2a Proof of Concept Study of Treatment of Chronic Fatigue Syndrome (CFS) With Iodinated Activated Charcoal (IodoCarb®)
Brief Title: Treatment of Chronic Fatigue Syndrome (CFS) With Iodinated Activated Charcoal (IodoCarb®)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PharmaLundensis AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PL1201
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IodoCarb (r) (Active Comparator): 3 g iodinated activated charcoal, IodoCarb(r), daily for 28 +-2 days.
  Interventions: Drug: IodoCarb (r)
- Placebo (Placebo Comparator): 3 g of non-iodinated activated charcoal daily for 28+-2 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IodoCarb (r) — Powder, 3 grams daily for 28+-2 days
  Arms: IodoCarb (r)
Other: Placebo — Non-iodinated activated charcoal 3 g daily for 28+-2 days
  Arms: Placebo

SUMMARY:
Chronic fatigue syndrome (CFS) is a devastating and complex disorder. People with CFS experience overwhelming fatigue and a host of other symptoms that are not improved by bed rest. Interestingly, many of the symptoms experienced by people with CFS are identical to symptoms caused by long-term low-level exposure to mercury, which is called micromercurialism.

This study will examine if the mercury binding substance IodoCarb(r) can improve the health of patients with CFS.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS, which is also sometimes called ME, Myalgic Encephalomyelitis) is a devastating and complex disorder. People with CFS experience overwhelming fatigue and a host of other symptoms that are not improved by bed rest and that can get worse after physical activity and mental exertion. They often function at a substantially lower level of activity than they were capable of before they became ill. Besides severe fatigue, other symptoms include muscle- and joint pain, impaired memory or mental concentration, insomnia, and post-exertion malaise lasting more than 24 hours. Often, CFS can persist for many years. Researchers have not yet identified what causes CFS, and there are no specific tests to diagnose CFS. The prevalence has been suggested to be around 1-2 %.

All humans are exposed to small amounts of mercury every day from the environment. It is well-known that exposure to mercury in small quantities for a long time can affect the psychic function, and cause severe fatigue, insomnia, lack of concentration and memory problems, which is called micromercurialism. It is also known that the sensitivity to the toxic effects by mercury differs greatly between people. Thus, it is quite possible that the small amount of mercury that humans are exposed to daily are sufficient to lead to micromercurialism symptoms in sensitive individuals. Therefore, the question arises if a reduction of the mercury content in the body of CFS patients can improve their symptoms and problems in daily life.

This study will examine if the mercury binding substance IodoCarb(r) can improve the health of patients with CFS.

This is a double blind placebo controlled parallel group study.

Patient population: 40 patients diagnosed with CFS will participate.

ELIGIBILITY:
Inclusion Criteria:

* Chronic fatigue syndrome
* 35-60 years old
* Male
* Female (not pregnant or breastfeeding, using adequate highly effective contraception consistently and correctly or >1 year post-menopausal or surgically sterile).

Exclusion Criteria:

* Iodine allergy
* abnormal thyroid function or other thyroid disease such as goiter
* severely reduced kidney function (Cystatin C > 1.5 mg/L)
* alcohol/drug abuse
* severe depression
* severe fibromyalgia
* severe cardio-vascular disease
* other severe disease, according to the clinical investigator
* participation in another ongoing clinical trial
* participation in drug trial the preceding 3 months

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire score | The QoL score during the last (fourth) treatment week is compared to the QoL score during the control week just prior to the treatment period.
  The QoL score during the last (fourth) treatment week is compared to the QoL score during the control week just prior to the treatment period. Results from patients receiving active substance will be compared to patients who received placebo.

SECONDARY OUTCOMES:
Use of psychotropic drugs | The intake of psychotropic drugs during the last (fourth) treatment week is compared to the intake during the control week just prior to the treatment period.
  The intake of psychotropic drugs (sedatives, anxiolytics or hypnotic drugs) during the last (fourth) treatment week is compared to the intake of psychotropic drugs during the control week just prior to the treatment period. Results from the IodoCarb group will be compared to results from the Placebo group.
Physical activity measured by a pedometer | The physical activity of patients during the last (fourth) treatment week is compared to the physical activity during the control week just prior to the treatment period.
  The physical activity of patients during the last (fourth) treatment week is compared to the physical activity during the control week just prior to the treatment period using a pedometer. Results from the IodoCarb group will be compared to results from the Placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Luts, MD, PhD, Principal Investigator — Probare i Lund AB
Locations (1):
- Probare i Lund AB, Lund, Sweden

REFERENCES:
- See also: The sponsor´s web site (in swedish) — http://www.pharmalundensis.se/